CLINICAL TRIAL: NCT03494361
Title: Evaluation of Dysphagia by 6-chnnel Surface Electromyography and Preliminary Study for Design 6-channel Electrical Stimulation
Brief Title: Evaluation of Dysphagia by 6-chnnel Surface Electromyography
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ju Seok Ryu, associate professor, Seoul National University Hospital
Other Study IDs: B-1604/344-003
Record Dates: First submitted 2018-04-02; First posted 2018-04-11 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Deglutition Disorders
Keywords: deglutition disorders; electromyography
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young normal group: normal participants below 60 years
- Old normal group: normal participants above 60 years

SUMMARY:
The natural process of aging affects a few very specific timing parameters such as swallow reaction time and hyoid one movement velocity.

Many swallow timing and bolus transit parameters appear to be unaffected by aging. We want to know the changes of kinematic variables according to the aging process.

First hypothesis: There are probably be a protection mechanism that blocks functional loss progressing to kinematic abnormality. Muscle activation sequence change (i.e duration or amplitude) of the oropharyngeal muscles play an important role.

Second hypothesis: Age-related differences in muscle activation patterns will also appear differently depending on the characteristics of swallowed food.

DETAILED DESCRIPTION:
Inclusion criteria

Inclusion criteria of healthy older adults : Age > 60, without dysphagia, comorbidity

Inclusion criteria of young control group

: Age < 60, without dysphagia, comorbidity

No prior history of swallowing difficulty or history of central nervous system disease, and none were taking medication that are known to affect swallowing.

Surface EMG was performed at bilateral suprahyoid, thyrohyoid, sternothyroid and pharyngeal constrictors. The latency of activation and termination was checked.

ELIGIBILITY:
Inclusion Criteria of old group

* Age > 60, without dysphagia, comorbidity

Inclusion Criteria of young control group

* Age < 60, without dysphagia, comorbidity

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy participants
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-07-04 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2017-11-21 (Actual)

PRIMARY OUTCOMES:
Latency | once at study, when patient enrolled
  the latency of muscular activation

SECONDARY OUTCOMES:
duration | once at study, when patient enrolled
  the contractile duration of evaluated muscles